CLINICAL TRIAL: NCT02594020
Title: Comparison of Different Methods of Enamel Preparation Before Pit and Fissure Sealants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 08-PP-09
Record Dates: First submitted 2013-06-04; First posted 2015-11-02 (Estimated); Last update posted 2016-04-25 (Estimated); Status verified 2015-09

CONDITIONS: Enamel Lesions; Dental Caries
Keywords: suspected caries; initial enamel lesions
MeSH Terms: conditions — Dental Caries | interventions — Air Abrasion, Dental

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- dental bur versus air abrasion (Other): 1 tooth prepared with air abrasion versus one prepared tooth with dental bur
  Interventions: Procedure: air abrasion; Procedure: dental bur
- sono abrasion versus dental bur (Other): 1 tooth prepared with sono abrasion ans 1 tooth prepared with dental bur
  Interventions: Procedure: sono abrasion; Procedure: dental bur
- air abrasion versus sono abrasion (Other): 1 tooth prepared with air abrasion versus 1 tooth prepared with sono abrasion
  Interventions: Procedure: air abrasion; Procedure: sono abrasion

INTERVENTIONS:
Procedure: air abrasion — already used intervention to prepare micro cavities of the dental to be treated by a photopolymerizable resin
  Arms: air abrasion versus sono abrasion; dental bur versus air abrasion
Procedure: sono abrasion — already used intervention to prepare micro cavities of the dental to be treated by a photopolymerizable resin
  Arms: air abrasion versus sono abrasion; sono abrasion versus dental bur
Procedure: dental bur — already used intervention to prepare micro cavities of the dental to be treated by a photopolymerizable resin
  Arms: dental bur versus air abrasion; sono abrasion versus dental bur

SUMMARY:
This study concerns the prevention of dental caries by sealing pits and fissures of permanent molars with a photopolymerizable resin. It must compare these three techniques Microdentisty (air abrasion, abrasion and sound using small cutters) usually used to prepare micro cavities in the enamel and / or the outer third of the dentin. These three commonly used techniques have never been compared by retaining as endpoint retention of sealant. These techniques are painless and do not require local anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* Affiliated with the Social Security
* Attendance at inspections
* Subject to high individual risk of caries
* Subjects with at least two pairs of molars and contralateral counterparts with the initial lesions of enamel (pits and fissures colored) or suspected of dentine caries (not highlighted by two clinical and radiographic examination usual)

Exclusion Criteria:

* Molar inaccessible, closed, sealed, or decayed (reaching the dentine

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Actual)
Dates: Start 2008-06; Primary Completion 2013-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
observation of quality of treatment | 2 years
  Compare enamel preparation techniques of air abrasion and sound abrasion technique enameloplasty (pits and fissures extended to the dental bur) the more conventionally used to identify the most effective as using endpoint retention of material sealing of pits and fissures.

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - CHU, Nice
  - APHP, Paris